CLINICAL TRIAL: NCT07144306
Title: AI-Driven Early Detection of Skin Cancer
Acronym: Skin Cancer
Status: Recruiting | Type: Observational
Sponsor: Nuvana Healthcare LTD (Industry)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 70148; 359904 (Other: IRAS)
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Skin Cancer Melanoma
Keywords: Skin Cancer; Melanoma; Early Detection; Artificial Intelligence; Dermatology; Digital Health
MeSH Terms: conditions — Melanoma; Skin Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with suspicious skin lesions undergoing AI-based image analysis and dermatologist confi
  Interventions: Diagnostic Test: Smartphone-based AI skin lesion analysis (NuvanaDx platform).

INTERVENTIONS:
Diagnostic Test: Smartphone-based AI skin lesion analysis (NuvanaDx platform). — Smartphone-based AI skin lesion analysis (NuvanaDx platform).

SUMMARY:
This study evaluates the feasibility and accuracy of an AI-powered mobile platform (NuvanaDx) for early detection of skin cancer, including melanoma, using smartphone-based imaging. The platform is designed to improve access to early diagnosis, reduce waiting times, and support triage into appropriate care pathways.

DETAILED DESCRIPTION:
The study will collect retrospective and prospective anonymized skin lesion images and metadata to validate the AI algorithm against dermatology-confirmed diagnoses. The aim is to determine sensitivity, specificity, and predictive value of the AI tool across diverse populations and skin tones. The study will also assess user experience, accessibility, and integration into clinical care pathways.

ELIGIBILITY:
Inclusion Criteria:

Adults (≥18 years) presenting with skin lesions suspicious for malignancy.

Ability to provide informed consent.

Exclusion Criteria:

Inability to provide informed consent.

Poor-quality images unsuitable for AI analysis.

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study Population Description: Individuals undergoing dermatology evaluation in UK clinics, supplemented by retrospective anonymized image datasets.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of AI tool compared with dermatologist-confirmed diagnosis | Time Frame: Up to 12 months
  Diagnostic Accuracy of AI tool compared with dermatologist-confirmed diagnosis
  Time Frame: Up to 12 months
  Measure: Sensitivity, specificity, and predictive values

CONTACTS AND LOCATIONS:
Overall Officials: Aryan Chaudhary,, Study Chair — Scientific Advisor / Co-Founder, Nuvana Healthcare
Locations (1):
- Nuvana Healthcare Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) that underlie the results of this study will be shared after de-identification. This will include anonymized image datasets of skin lesions (with corresponding dermatology-confirmed diagnoses), demographic variables (age, sex), and relevant clinical outcomes. No personally identifiable information (PII) will be shared. Data will be made available for the purpose of secondary analysis, validation studies, and meta-analyses in the field of dermatology, oncology, and digital health.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified IPD and supporting information will be available beginning 6 months after study completion (anticipated June 2027). Data will remain available for at least 5 years (until December 2032), after which access will be reviewed and may be extended based on scientific demand.
Access Criteria: Access will be granted to qualified researchers affiliated with academic institutions, non-profit organizations, or healthcare systems, upon submission of a research proposal that aligns with the study's objectives. Proposals will be reviewed by Nuvana Healthcare's Scientific Advisory Board. Data will be shared under a data use agreement (DUA) to ensure confidentiality and compliance with ethical standards. Access will be provided through a secure, password-protected platform, with no download of raw datasets permitted unless explicitly approved.
URL: https://www.nuvana.co.uk